CLINICAL TRIAL: NCT02601976
Title: Response Evaluation of Peginterferon Alfa-2a 180µg 20kDa (Unipeg®) Plus Ribavirin (Ribazole®) in Treatment naïve Pakistani Population With Chronic Hepatitis C Infection
Brief Title: Evaluation of Unipeg® for Response and Ongoing Safety in Pakistani Population
Acronym: EUROP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Collaborators: Dimension Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETZ-UNIP- 4010810
Record Dates: First submitted 2015-11-02; First posted 2015-11-11 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
Keywords: PegInterferon alpha-2a; Ribavirin; Hepatitis C Virus; Sustained Virological Response; End of Treatment Response; Unipeg; Ribazole
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin; alpha-ribazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PegInterferon alfa-2a and Ribavirin (Experimental): PegInterferon alfa-2a subcutaneously once weekly Ribavirin administered orally according to the body weight
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a — PegInterferon alfa-2a 180mcg 20kDa administered subcutaneously once weekly for 24 weeks in genotype 3 and for 48 weeks in genotype 1 patients.
  Other Names: Unipeg
Drug: Ribavirin — Ribavirin administered orally in a divided daily dose according to body weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribazole

SUMMARY:
Hepatitis C is a global problem, prevalent in developed as well as in the developing countries. New treatment regimens using PegInterferon in combination with ribavirin has led to improved sustained viral response rates for some genotypes. A single arm, open labeled, multicentre trial was conducted to evaluate the response rate and safety of PegInterferon alfa-2a (Unipeg®) plus ribavirin (Ribazole®) for the treatment of patients with chronic hepatitis C infection. RVR at 4 weeks, ETR at 24 weeks for genotype 3 and at 48 weeks for genotype 1 patients and SVR was determined at 24 weeks after completion of treatment. Quality of life at baseline and at follow-up visits were determined using SF-36.

DETAILED DESCRIPTION:
A multicenter, phase IV, open labeled, single arm study was conducted. Total 110 patients were screened for recruitment. Out of which 67 subjects met the inclusion criteria, 3 failed to give the informed consent and were excluded. The final sample size of the study was 64 patients. The duration of study was August 2010 to September 2013. Peginterferon alfa-2a 180µg 20kDa (Unipeg®) solution for injection was administered as single dose sub-cutaneous once weekly for 24 weeks to patients with genotype 3 and 48 weeks in patients with genotype 1 at the site of recruitment. Ribavirin (Ribazole) orally were given in divided daily dose according to body weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg). Quality of life related Physical Component Score (PCS) & Mental Component Score (MCS) were measured through Health-Related Quality of Life (HRQOL) Questionnaire (SF-36). The SF-36 questionnaire was completed for all patients during their evaluations before treatment, at 4 weeks, at the end of treatment and at 24 weeks after completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed consent
2. Treatment naïve patients
3. Serological evidence of hepatitis C infection by an anti-HCV antibody test
4. HCV positive by PCR
5. Genotype 1,2 and 3
6. BMI 20-28
7. Participants were the resident of city where he /she enrolled at their respective centre
8. No evidence of liver cirrhosis
9. No other significant hepatic or systemic disease
10. No evidence of hepatic encephalopathy
11. Normal thyroid functions (By testing TSH)
12. Adequate bone marrow, liver and renal functions test

    * Hematology: ANC≥1,000/mm3, Platelet count ≥100,000 mm3, Hemoglobin≥11.0g/dl in female and ≥ 12.0 g/dl in male
    * Blood Chemistry: Total Bilirubin≤2.0mg/dl, AST and ALT <3 times normal
    * Creatinine Clearance >50 ml/min
    * Proteinuria: ≤ 0.5 g per 24h.
    * Prothrombin Time or partial-thromboplastin time if ≤1.5 times the upper limit of the normal range.

Exclusion Criteria:

1. Unable to give consent
2. Prior treatment for Hepatitis C
3. Co-infection with HBV and HCV
4. Obesity
5. Iron overload
6. Other Genotypes e.g. 4, 5, 6 with their sub-types
7. Pregnant and lactating women
8. History of medical condition associated with chronic liver disease other than CHC (e.g. hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposure)
9. Uncontrolled Hypertension
10. Uncontrolled Diabetes
11. Severe Depression
12. Clinically significant cardio-vascular disease
13. Symptomatic peripheral vascular disease
14. Oral or parenteral anticoagulants or anti platelet agents
15. History of systemic anti-viral therapy at least three months prior to first dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Khawar Mehdi, MD, Study Director — Getz Pharma Pakistan

REFERENCES:
- [Background] Chander G, Sulkowski MS, Jenckes MW, Torbenson MS, Herlong HF, Bass EB, Gebo KA. Treatment of chronic hepatitis C: a systematic review. Hepatology. 2002 Nov;36(5 Suppl 1):S135-44. doi: 10.1053/jhep.2002.37146. PMID 12407587
- [Background] Abbas Z, Jeswani NL, Kakepoto GN, Islam M, Mehdi K, Jafri W. Prevalence and mode of spread of hepatitis B and C in rural Sindh, Pakistan. Trop Gastroenterol. 2008 Oct-Dec;29(4):210-6. PMID 19323090
- [Background] Ali SA, Donahue RM, Qureshi H, Vermund SH. Hepatitis B and hepatitis C in Pakistan: prevalence and risk factors. Int J Infect Dis. 2009 Jan;13(1):9-19. doi: 10.1016/j.ijid.2008.06.019. Epub 2008 Oct 2. PMID 18835208
- [Background] European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. No abstract available. PMID 25911336
- [Background] Idrees M, Riazuddin S. Frequency distribution of hepatitis C virus genotypes in different geographical regions of Pakistan and their possible routes of transmission. BMC Infect Dis. 2008 May 23;8:69. doi: 10.1186/1471-2334-8-69. PMID 18498666
- [Background] Hadziyannis SJ, Sette H Jr, Morgan TR, Balan V, Diago M, Marcellin P, Ramadori G, Bodenheimer H Jr, Bernstein D, Rizzetto M, Zeuzem S, Pockros PJ, Lin A, Ackrill AM; PEGASYS International Study Group. Peginterferon-alpha2a and ribavirin combination therapy in chronic hepatitis C: a randomized study of treatment duration and ribavirin dose. Ann Intern Med. 2004 Mar 2;140(5):346-55. doi: 10.7326/0003-4819-140-5-200403020-00010. PMID 14996676
- [Background] Ahmad, T., R. Ahsan, and G. Saba. Evaluation of Safety and Pharmacokinetic Behavior of Unipeg® in Healthy Human Volunteers. Journal of Pharmacy and Nutrition Sciences 2014;4.3:220-227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
Age, Customized [Mean (Standard Deviation); unit: participants]
  Count | 35.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Count: Female | 28
  Count: Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 64
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Pakistan | 64
Number of HCV Patients confirmed through Polymerase Chain Reaction [Number; unit: participants] — Patients sent for Polymerase Chain Reaction (PCR) Lab investigation and those were selected who had positive PCR.
  participants | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virological Response (SVR)
Description: To determine the SVR at 24 weeks after completion of treatment, among those who achieved ETR
Time Frame: Post treatment Week 24
Population: Among those who achieved ETR (i.e. 56 participants) were eligible for SVR analysis after 24 weeks of post treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 56
Participants | 49

2. Primary Outcome: Number of Participants With End Treatment Response
Description: To determine the End Treatment Response (ETR) rate of all patients treated with PegInterferon alfa-2a plus Ribavirin
Time Frame: Upto 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
Participants | 56

3. Secondary Outcome: Number of Participants Who Reported Adverse Events
Description: To determine the number of patients treated with PegInterferon Alfa-2a plus Ribavirin who experience any adverse drug reaction. All ADR are reported as per patient information leaflet
Time Frame: Upto 48 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
Participants | 10

4. Other Pre Specified Outcome: Number of Participants With Rapid Virological Response (RVR)
Description: To evaluate the Rapid Virological Response (RVR) of all patients treated with PegInterferon Alfa-2a plus Ribavirin at 4 weeks of treatment
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
Participants | 48

5. Other Pre Specified Outcome: Mean of Physical Component Score & Mental Component Score to Determine Quality of Life
Description: To determine and compare the changes in quality of life (QOL) from baseline to end of the treatment. Health-Related Quality of Life (HRQOL) Questionnaire (SF-36) was used to measure the quality of life. The SF-36 is a widely used questionnaire, and consists of 36 questions measuring eight concepts: Physical Function (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Function (SF), Role Emotional (RE), and Mental Health (MH). The scoring of the SF-36 questionnaire in our study was conducted upon a 0-100 scale, with higher scores reflecting better health status.
Time Frame: Upto 48 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PegInterferon Alfa-2a and Ribavirin
Number analyzed (Participants) | 64
score on a scale
  Physical Component Score | 50.62 (8.22)
  Mental Component Score | 54.89 (9.61)

ADVERSE EVENTS:
Arm/Group | PegInterferon Alfa-2a and Ribavirin
All-Cause Mortality (participants affected / at risk) | 10/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 10/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PegInterferon Alfa-2a and Ribavirin (N=64)
Body Pain (General disorders) | 5
Rashes (Immune system disorders) | 2
Epigastric Pain (Gastrointestinal disorders) | 2
Flu (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes